CLINICAL TRIAL: NCT00224679
Title: Prospective Study on Aspirin Efficacy in Reducing Colorectal Adenoma Recurrence
Brief Title: APACC Study:Prospective Study on Aspirin Efficacy in Reducing Colorectal Adenoma Recurrence
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Société Nationale Française de Gastroentérologie (Other); Ministry of Health, France (Other Government); Sanofi-Synthelabo (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AOM 95176; P951202; RAF 95176
Record Dates: First submitted 2005-09-19; First posted 2005-09-23 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2006-09

CONDITIONS: Colon Adenomas
Keywords: Colon cancer; Aspirin; Adenomas; Prevention
MeSH Terms: conditions — Colonic Neoplasms; Adenoma | interventions — Aspirin

INTERVENTIONS:
Drug: Aspirin

SUMMARY:
Experimental and epidemiologic studies have suggested that aspirin intake reduces the risk for colorectal cancer. In the APACC study we randomly assigned 291 patients to daily Aspirin or Placebo for 4 years. However, the available data are not sufficient to serve as the basis for firm recommendations

DETAILED DESCRIPTION:
The APACC Study is a prospected, randomized, double-blind, placebo-controlled multicentre clinical trial design to test the efficacy of regular low-dose aspirin administration in reducing the recurrence rate of colorectal adenomatous polyps. The study involved 49 gastroenterology centers from various parts of France. Patients were eligible if they had either at least 3 adenomas irrespective of size, or at least one measuring 6mm in diameter or more histologically confirmed colorectal adenomatous polyp by the local pathologist, and 2 independent pathologists, underwent a complete colonoscopy with polypectomy and were then confirmed free of polyps, were aged between 18 and 75 years at recruitment, and were be able to conform to the protocol during the study period. During a 4-week run-in period before enrolment, all subjects took 300 mg aspirin per day to test tolerance and compliance with the treatment. They were then randomized to either of the following three groups: placebo, aspirin as acetylsalicylate of lysine 160 mg/day or aspirin as acetylsalicylate of lysine 300 mg/day. Information on compliance, tolerance of the treatment and concomitant disease is obtained at regular clinical visits every 4 months. Informations on factors such as smocking habits, previous medical history was recorded at enrollment. The primary outcomes were defined as the proportion of subjects in whom at least one new adenoma was detected, and the adenomatous polyp burden calculated as the sum of the diameters of these adenomas at the follow-up colonoscopy 1 and 4 years after enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Patients are aged between 18 and 75 years At least 3 adenomas irrespective size or at least one measuring 6mm or more All subjects had a clean colon at the study entry

Exclusion Criteria:

* No personal history of colon cancer, no inflammatory bowel disease, no familial adenomatous polyposis, no regular use of aspirin

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 1997-03; Study Completion 1999-03

PRIMARY OUTCOMES:
Is daily soluble aspirin associated with a reduction in the risk for recurrent adenomas at 1 and 4 years after starting treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Stanislas CHAUSSADE, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital COCHIN Service d'Hépato-Gastro-Entérologie, Paris, Île-de-France Region, France

REFERENCES:
- [Background] Benamouzig R, Deyra J, Martin A, Girard B, Jullian E, Piednoir B, Couturier D, Coste T, Little J, Chaussade S. Daily soluble aspirin and prevention of colorectal adenoma recurrence: one-year results of the APACC trial. Gastroenterology. 2003 Aug;125(2):328-36. doi: 10.1016/s0016-5085(03)00887-4. PMID 12891533
- [Derived] Benamouzig R, Uzzan B, Deyra J, Martin A, Girard B, Little J, Chaussade S; Association pour la Prevention par l'Aspirine du Cancer Colorectal Study Group (APACC). Prevention by daily soluble aspirin of colorectal adenoma recurrence: 4-year results of the APACC randomised trial. Gut. 2012 Feb;61(2):255-61. doi: 10.1136/gutjnl-2011-300113. Epub 2011 Sep 2. PMID 21890814